CLINICAL TRIAL: NCT07024693
Title: A Phase 2, Multicenter, Open-Label Study to Assess the Pharmacodynamics, Safety, and Tolerability of DT-168 Ophthalmic Solution in Patients With Fuchs Endothelial Corneal Dystrophy Undergoing Keratoplasty
Brief Title: DT-168 in Keratoplasty Patients With Fuchs Endothelial Corneal Dystrophy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Design Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DTX-168-201
Record Dates: First submitted 2025-05-20; First posted 2025-06-17 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Fuchs Endothelial Corneal Dystrophy; Fuchs
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Active (Experimental): Drug: DT-168
  Interventions: Drug: DT-168

INTERVENTIONS:
Drug: DT-168 — Active

SUMMARY:
The purpose of this study is to evaluate the pharmacodynamics, safety, and tolerability of DT-168 Ophthalmic Solution in pre-keratoplasty patients with Fuchs endothelial corneal dystrophy.

ELIGIBILITY:
Inclusion Criteria:

* Participant is scheduled to undergo a keratoplasty for management of FECD independent of this study.
* ≥30 years of age (inclusive).
* Documented diagnosis of FECD in the study eligible eye.
* Confirmation of positive TCF4 allele 18.1 CTG expansion in at least one allele.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Any ocular or medical condition in the study eligible eye which is clinically significant or would confound study results or data interpretation.
* Any clinically significant medical, nonmedical, and psychiatric disorders that could put the participant at higher risk for participation in the study, impair the participant's ability to participate in the study, or interfere with interpretation of the participant's study results, in the opinion of the investigator.
* Concurrent or anticipated need for treatment for FECD, eg, Muro 128 (2% or 5%) during the course of the study in the study eye. Provided the subject undergoes a washout of Muro drops for at least 24 hours prior to the Baseline Visit, they will not be excluded.
* Concurrent or anticipated use of topical corticosteroids in the study eye.
* Concurrent use with Rhopressa®, Rocklatan®, or any other ocular Rho Kinase inhibitor.
* Known contraindication, allergy, or hypersensitivity to any of the treatments, anesthetics, or diagnostic agents or components thereof which may be used during the study.
* Use of contact lenses in the study eye within 7 days prior to the Baseline Visit or planned use during the study.
* Recent (within 30 days of the Screening Visit) or ongoing participation in any other investigational interventional clinical study.
* Female participant is pregnant, planning a pregnancy, or breast-feeding.
* Participant is unwilling to comply with the contraceptive requirements, as per protocol.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
FECD Biomarkers: Splicing Panel | Perioperative
  Assessment of DT-168 on splicing patterns in genes that are known to be disrupted in FECD.

SECONDARY OUTCOMES:
Safety and Tolerability | Through study completion, an average of 4 weeks.
  Frequency of treatment-emergent adverse events

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - DTX-168-201 Study Site, Indianapolis, Indiana
  - DTX-168-201 Study Site, Grand Rapids, Michigan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.designtx.com